CLINICAL TRIAL: NCT06390436
Title: Therapeutic Drug Monitoring-baSed adalimuMab De-escalatiOn in nOn-infecTious cHronic Uveitis: an Open-label, Non-inferiority, Randomised Clinical Trial
Brief Title: Therapeutic Drug Monitoring-baSed adalimuMab De-escalatiOn in nOn-infecTious cHronic Uveitis
Acronym: SMOOTH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23PH187; 2023-509733-39-00 (Other: CTIS)
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Uveitis; Chronic Disease
Keywords: Adalimumab; Uveitis; Therapeutic drug monitoring
MeSH Terms: conditions — Uveitis; Chronic Disease | interventions — Blood Specimen Collection; Adalimumab

STUDY DESIGN:
Intervention Model Description: SMOOTH is a multicenter, randomized, controlled, parallel-group, blinded end-point trial (Prospective Randomised Open, Blinded End-point, PROBE) designed to demonstrate the superiority of a TDM-based strategy of therapeutic de-escalation via the spacing of ADA administrations versus a conventional ADA-based therapeutic strategy.
Who Masked: Investigator
Masking Description: The primary endpoint will be assessed by blinding the allocated treatment group to investigator.
  Thus, ophthalmological response will be assessed in a standardised manner by an ophthalmologist, blinded to the treatment strategy. The occurrence of infections will also be assessed in a manner blinded to the by an independent adjudication committee.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm : conventional strategy (Active Comparator): At W0, ADA administration will be continued every 14 days. At W24, the control arm will continue to receive ADA every 14 days regardless of serum ADA concentration.
  Interventions: Diagnostic Test: Blood sample; Drug: Adalimumab Injection
- Arm 2: Interventional arm : adalimumab dose spacing strategy (Experimental): At W0, if the serum ADA concentration is ≥ 8 μg/mL, ADA administration will be spaced every 21 days. At W24, if the ADA concentration is < 3.3 μg/mL (having a serum ADA concentration above this threshold was associated with a complete therapeutic response according to one study), administrations will be repeated every 14 days. If the ADA concentration is ≥ 3.3 and < 8μg/mL, administrations will be left every 21 days. If ADA concentration is still ≥8μg/mL, ADA administrations will be spaced every 28 days.
  Interventions: Diagnostic Test: Blood sample; Drug: Adalimumab Injection

INTERVENTIONS:
Diagnostic Test: Blood sample — A blood sample will be taken, in addition to blood samples taken for the usual follow-up, with 4 dry tubes for the determination of ADA and anti-ADA antibodies and for bio-collection.
Drug: Adalimumab Injection — Adalimumab Injection

SUMMARY:
Uveitis and its complications are thought to account for 10 to 15% of preventable blindness in Western countries. The diagnosis of chronic non-infectious uveitis (CNUI) can be made after exclusion of pseudo uveitis or infectious uveitis, in the case of any persistent uveitis or uveitis with frequent relapses occurring less than 3 months after cessation of treatment. Adalimumab (ADA), an anti-TNFα monoclonal antibody, has marketing authorization and is widely used in the treatment of UCNI as a relay to corticosteroids. The use of ADA has been optimized, in particular through Therapeutic Drug Monitoring (TDM), based on the determination of serum ADA levels and anti-ADA antibodies. Recently, an article showed that a strategy of spacing ADA administrations in RA patients with concentrations >8 μg/mL was not inferior to standard.

DETAILED DESCRIPTION:
There is currently no formal recommendation for spacing ADA administration in patients with chronic noninfectious uveitis, but promising data from a recent retrospective study conducted by the Croix-Rousse team, led to the proposal of a decision support algorithm. Following the example of what has been shown in rheumatoid arthritis, the investigators propose to compare a strategy of spacing ADA administrations in patients with a satisfactory clinical response associated with high serum ADA concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Informed and having signed the study consent form
* Age ≥ 18 years
* NICU according to the Standardization of Uveitis Nomenclature (SUN) criteria
* Complete ophthalmological response for ≥ 48 weeks (96 weeks for uveitis related to Behçet's disease), all treatments combined
* On ADA 40mg / 14 days for ≥ 24 weeks (i.e. achievement of the steady state for ADA concentrations)
* Not having received systemic corticosteroid therapy for ≥ 12 weeks

Exclusion Criteria:

* Inability or refusal to understand and/or sign the informed consent form to participate in the study.
* Inability and/or refusal to carry out the follow-up examinations required for the study.
* Modification of any background immunomodulatory treatment (e.g. methotrexate, hydroxychloroquine, mycophenolate, etc.) associated with ADA, during the 12 weeks prior to inclusion.
* Uveitis suspected or proven to be of infectious origin
* Planned surgery (or other foreseeable medical event) requiring discontinuation of ADA for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Maintenance of a complete ophthalmological response at 48 weeks | Week 48
  Number of patient with complete ophthalmological response. Ophtalmological response is defined as number of patient with, in both eyes, absence of inflammatory lesions (0 = absence) AND a cellular grade of the anterior chamber and vitreous ≤ 0.5+.
Infection | Week 48
  Number of infection during follow-up for up to 48 weeks. Any suspected infectious event will have to be validated by a healthcare professional based on the presence of suggestive clinical signs (purulent sputum, fever ≥38°C, inflammatory syndrome, positive microbiological examination, etc.) via dedicated forms and validated by an adjudication committee.

SECONDARY OUTCOMES:
Maintenance of a complete ophthalmological response at 12 weeks | Weeks 12
  Number of patient with complete ophthalmological response. Ophtalmological response is defined as number of patient with, in both eyes, absence of inflammatory lesions (0 = absence) AND a cellular grade of the anterior chamber and vitreous ≤ 0.5+.
Maintenance of a complete ophthalmological response at 24 weeks | Weeks 24
  Number of patient with complete ophthalmological response. Ophtalmological response is defined as number of patient with, in both eyes, absence of inflammatory lesions (0 = absence) AND a cellular grade of the anterior chamber and vitreous ≤ 0.5+.
Maintenance of a complete ophthalmological response at 36 weeks | Weeks 36
  Number of patient with complete ophthalmological response. Ophtalmological response is defined as number of patient with, in both eyes, absence of inflammatory lesions (0 = absence) AND a cellular grade of the anterior chamber and vitreous ≤ 0.5+.
Infection | Week 12
  Number of infection during follow-up for up to 12 weeks. Any suspected infectious event will have to be validated by a healthcare professional based on the presence of suggestive clinical signs (purulent sputum, fever ≥38°C, inflammatory syndrome, positive microbiological examination, etc.) via dedicated forms and validated by an adjudication committee.
Infection | Week 24
  Number of infection during follow-up for up to 24 weeks. Any suspected infectious event will have to be validated by a healthcare professional based on the presence of suggestive clinical signs (purulent sputum, fever ≥38°C, inflammatory syndrome, positive microbiological examination, etc.) via dedicated forms and validated by an adjudication committee.
Infection | Week 36
  Number of infection during follow-up for up to 36 weeks. Any suspected infectious event will have to be validated by a healthcare professional based on the presence of suggestive clinical signs (purulent sputum, fever ≥38°C, inflammatory syndrome, positive microbiological examination, etc.) via dedicated forms and validated by an adjudication committee.
Anti-ADA antibody positivity | Weeks 12
  Anti-ADA antibody positivity by a "drug sensible" test (i-Tracker anti-ADA) in μg/mL
Anti-ADA antibody positivity | Weeks 24
  Anti-ADA antibody positivity by a "drug sensible" test (i-Tracker anti-ADA) in μg/mL
Anti-ADA antibody positivity | Weeks 36
  Anti-ADA antibody positivity by a "drug sensible" test (i-Tracker anti-ADA) in μg/mL
Anti-ADA antibody positivity | Weeks 48
  Anti-ADA antibody positivity by a "drug sensible" test (i-Tracker anti-ADA) in μg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Lucile GRANGE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (11):
- France (11):
  - CH Avignon, Avignon
  - Chu Montpied, Clermont-Ferrand
  - CHU Grenoble Alpes, Grenoble
  - CH Le Puy-en-Velay, Le Puy-en-Velay
  - Hôpital de la Croix Rousse, Lyon
  - HCL - Hôpital Edouard Herriot, Lyon
  - CHU MONTPELLIER - Hôpital Saint-Eloi, Montpellier
  - APHP - Centre hospitalier national des Quinze-Vingts, Paris
  - APHP - Hôpital Pitié-Salpétrière, Paris
  - APHP - Hôpital Cochin, Paris
  - Chu de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No